CLINICAL TRIAL: NCT06321627
Title: Radiosensitivity of HPV-related Tumors: Towards a Genomic Approach - ICARUS Project
Brief Title: Radiosensitivity of HPV-related Tumors: Towards a Genomic Approach
Acronym: ICARUS
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1811
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: HPV-Related Carcinoma
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with HPV-related tumors: Patients with HPV-related tumors of the oropharynx, cervix, and anus
  Interventions: Radiation: Radiation therapy as curative treatment

INTERVENTIONS:
Radiation: Radiation therapy as curative treatment — Radiation therapy as curative treatment (exclusive, post-operative, with or without chemotherapy) for HPV-related squamous cell carcinomas of the oropharynx, uterine cervix, and anus

SUMMARY:
The purpose of this study is therefore to analyze the genomic profiles of prognosis and radiosensitivity of Human Papilloma Virus (HPV) related tumors from different body sites (oropharynx, uterine cervix, and anus), considering them as a unified entity regardless of the site of origin within the body.

DETAILED DESCRIPTION:
The present study (ICARUS - genomIC RAdiosensitivity viRUS) involves the collection of data (retrospective and prospective) from an extensive cohort of patients with HPV-related tumors of the oropharynx, cervix, and anus.

The aim is to:

1. investigate the role of Cl2 in non-oropharyngeal HPV-related tumors, and
2. compare the Radiation Sensitivity Index (RSI) values of HPV-related tumors in patients who responded to radiotherapy (responders) with those of patients with radioresistant tumors (non-responders).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old)
* Diagnosis of HPV-related squamous cell carcinomas of the oropharynx, uterine cervix, and anus
* Curative intent radiation therapy (exclusive, post-operative, with or without chemotherapy)
* Availability of pre-radiation therapy biopsy sample
* No diagnosis of solid neoplasms and/or hematologic malignancies in the previous 5 years
* Possibility of retrospective and prospective data collection and anonymous submission to the referring center of clinical data related to the patient, pathology, and treatment characteristics (including radiation treatment plan in RT.dose format)
* Ability to obtain written informed consent for the use of data anonymously for research purposes

Exclusion Criteria:

* Patients undergoing surgical treatment
* Patients with local and/or locoregional recurrence
* Patients with synchronous distant metastases at diagnosis
* Patients previously treated with oncologic therapies for tumors of the same anatomical site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HPV-positive tumors of the oropharynx, uterine cervix, and anus
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 5 years
  Number of patients with a recurrence (local or distant) after 5 years

SECONDARY OUTCOMES:
Genetic patterns of radiosensitivity | 1 year
  The biopsy samples from patients included in the database will be collected for the validation analyses of RadioSensitivity Index (RSI). The calculation of RSI will be performed using a panel of 10 genes extracted from the tumor biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Alterio, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy